CLINICAL TRIAL: NCT02219204
Title: Randomised Research Comparing Acupuncture, Herbal Treatment and Artificial Tear Eye Drops in Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R1142/44/2014; 2014/398/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-02

CONDITIONS: Dry Eye
Keywords: Acupuncture; Herbal treatment
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture treatment (Active Comparator): This will be performed twice weekly for 30 days. There will be 8 sessions of acupuncture treatments in total.
  The needles to be use around the eyes will have the dimensions of 0.25 (diameter) x 13mm (length), while 0.25 x 25mm needles will be used behind the ear (feng chi) and 0.30 X 25mm needles on the upper and lower limbs. These needles will remain in the points for 20 minutes. The depth of penetration will be about 1-2 mm.
  Interventions: Procedure: Acupuncture
- Herbal treatment (Active Comparator): This formulation is called qi ju gan lu yin or Lycium berry, a chrysanthemum beverage. This is a modified version of "qi ju di huang wan" published previously. The senior TCM collaborator, Prof Wei QP has made this modification in order to treat the dry eye patients with "lung-kidney yin deficiency".
  Interventions: Other: Herbal treatment
- Eye drops (No Intervention)

INTERVENTIONS:
Procedure: Acupuncture
  Arms: Acupuncture treatment
Other: Herbal treatment
  Arms: Herbal treatment

SUMMARY:
Dry eye is a major, common medical condition with significant health and economic burden in Singapore and worldwide. It is a holistic problem affected by living habits, nutrition and underlying systemic disease, inducing a significant decrease in quality-of-life. The hallmark of this disease is raised tear osmolarity and inflammation. There is no definitive cure for this condition, as treatment in the form of lubricants is only symptomatic and treatment with cyclosporine eyedrops is expensive and may not be well tolerated.

Following the rise in international interest in complementary medicine, randomized-controlled studies in dry eye using Traditional Chinese Medicine (TCM) have been published, with mixed results. However, the major limitation of these studies is the lack of objective assessment for inflammation.

We propose to collaborate with an academically-trained Singapore TCM physician who has conducted dry eye trials, and synergistically exploit the existing state-of-the-art dry eye monitoring technologies available at Singapore Eye Research Institute (SERI). This proposal is cost-effective, building on previous government grants and expertise to provide definitive scientific evidence on the efficacy and safety of TCM in dry eye. SERI has an international reputation for interventional studies, and the PI has a good academic relationship with the above TCM physician. We propose to screen, recruit and treat 150 patients with a herbal preparation and acupuncture, and evaluate over 4 weeks in a randomized-controlled study. Tests to be performed will include tear imaging and osmolarity, as well as protein and cytokine assays.

Singapore is uniquely positioned at the crossroads of the East and the West to take the lead in this field. Given that there is an increasing patient interest in holistic care in Singapore and the rise of scientifically trained TCM practitioners, a study like this one is very timely, and will have tremendous impact to healthcare delivery in Singapore.

DETAILED DESCRIPTION:
Dry eye is a major, common medical condition with significant health burden in Singapore and worldwide. As much as one third of the adult population in Asian countries are affected by dry eye. It has been shown that dry eye affects quality of life, including the performing of daily activities such as reading and driving a car. Moderate severity of dry eye affects some patients like moderate angina. The direct and indirect cost of treating dry eye is high and increasing. For example, it costs individuals about US$800 per year to treat dry eye, but the cost to society for managing such a patient is US$12000 per year. (1-29)

Dry eye is a holistic problem affected by living habits such as working long hours on the computer and in a dry, air-conditioned environment. It is also associated with poor nutrition and intake of dietary supplements such as omega-3 and omega-6 fatty acids may help to treat dry eye. Dry eye is also a systemic immune mediated disease, and aggravated by those with autoimmune Sjögren's syndrome, rheumatoid arthritis, thyroid disease, systemic lupus erythematosis, Steven Johnson syndrome and chronic graft versus host disease.

In a recent international workshop, international experts in dry eye agree that the hallmark of this disease is raised tear osmolarity and ocular surface inflammation. Traditionally, dry eye is diagnosed by a reduced Schirmer's test and/or reduced tear break up time or the presence of dry eye symptoms. In addition to these traditional tests, it would be advantageous to incorporate measurements of osmolarity and inflammation in clinical studies. There is no definitive cure for this condition, as treatment in the form of lubricants is only symptomatic and treatment with cyclosporine eye drops is expensive and may not be well tolerated. Treatment with steroids can be effective but associated with adverse effects such as sight threatening glaucoma. In summary there is a definite medical need for alternative therapies in dry eye.

Traditional Chinese Medicine (TCM) is involved in restoring the natural balance of the body, which results in disease like dry eye when this is disturbed. In TCM philosophy, dry eye may result from syndromes such as yin deficiency in the liver or kidney. Modalities such as acupuncture or herbs can be used judiciously to restore the balance in specific patients.

Recently there have been randomized controlled studies in dry eye using acupuncture and herbs, with mixed results, refer to attachment (Table 1). The major limitation of these studies is that objective tear film evaluation such as tear osmolarity, and tear cytokines and proteins, which are indicative of ocular surface inflammation, have not been evaluated. In addition, some studies suffer from lack of proper controls or randomization.

If the mainstream practitioners of evidence based medicine are convinced that TCM can fundamentally alter the pathological processes in dry eye, they will be more receptive to this form of treatment. At the same time, regulatory bodies need to be reassured that TCM is safe in dry eye, so that more education and promotion of such treatment can benefit more people.

The PI runs a dry eye clinic twice a week at the Singapore National Eye Centre since 2006. He is aware that many dry eye patients in Singapore have experienced a host of more conventional therapies and are eager to attempt alternative forms of therapy. This trend towards TCM and holistic medicine will continue regardless of the attitudes of 'western' medical practitioners. This study, when completed, will present an opportunity for bridging the gaps between the two health care communities who do not normally interact. Since latest scientific tools in terms of protein science and imaging will be employed in the study, it will definitely increase the evidence based medicine for TCM in the dry eye field.

The PI has published 67 peer reviewed papers in dry eyes and related ocular surface processes, including review articles,(30-34) international expert panel report,(35) epidemiological studies,(36-37) PI initiated and industry sponsored interventional drugs including randomized controlled drug trials.(38-40) In one pharmacy in Singapore alone, the cost of dry eye medications amounted to US$1.5 million in one year.(3) He has also found in an epidemiological study in Singapore people that dry eye impairs visual associated function related activities of daily living.(41) He established the only dedicated dry eye service in the region and has produced many papers relating to the assessment of these patients,(42-46) including one that found dry eye being related to the amount exposure to stressful activities and conditions.(46) The PI has experience in the biochemical evaluation of patient tears and materials in dry eye(47-51) and clinical imaging related to dry eye.(52-54) Lastly, he has also appeared in mass media educational articles including press releases and articles/talks for layperson and general practitioners.

A survey was conducted among registered TCM practitioners in Singapore and published in a peer reviewed journal.(55) This showed that a significant proportion of these institutional practitioners are keen to practice in dry eye. This study was also chosen to be presented as an oral presentation at the 10th Asean Congress of TCM cum 3rd Asia Advanced Forum on Acupuncture and Moxibustion. At the same time, the full article has been translated into Chinese in the congress proceedings page 192-197 to appeal to the audience of TCM physicians. The PI has also participated in discussion on data analysis in TCM trials. (56-57) In addition, acupuncture in rabbits had shown to induce changed in tear proteins, although this has not been evaluated in humans. (58)

1. HYPOTHESIS AND OBJECTIVES

   The overall hypothesis is that traditional Chinese medicine modalities of acupuncture and herbs can improve the symptoms and signs of dry eye, and objectively, these improvements are associated with reduction of tear osmolarity and reduction of inflammatory markers such as tear cytokines and proinflammatory proteins. There is also a long term objective of integrating TCM and mainstream medical care and having a cost-effective approach to eye disease.

   Primary outcome:

   • Change in SPEED score (Week4-Week0)

   Secondary outcomes:
   * Change in Tear Evaporimetry
   * Change in TCM score (Lung-Kidney Yin deficiency)
   * Change in NIBUT
   * Change in Schirmers I
   * Change in Corneal fluorescein staining (5 zones)
   * Change in Tear osmolarity
   * Change in Tear meniscus height
   * Change in Tear protein/ cytokine levels

   1.1 Primary Objectives

   We aim to show that dry eye patients treated with acupuncture is efficacious (can improve symptoms and signs of dry eye) and safe (no ocular and systemic side effects).

   1.2 Secondary Objectives

   We aim to show that dry eye patients treated with a herbal preparation is efficacious (can result in reduction of symptoms and signs of dry eye) and safe (no ocular and systemic side effects).

   We also aim to show that objective, definitive hallmarks of dry eye disease, ie. Tear osmolarity and surrogates of ocular surface inflammation, such as tear cytokines and proinflammatory proteins, are reduced after treatment by acupuncture and herbal treatment, compared to control.

   1.3 Potential Risks and Benefits: 1.3.1 Potential Risks We will anticipate minimal risk and discomfort involve in this study.
   * It is possible that eyelid bruising and swelling may occur from acupuncture needles
   * Some slight discomfort from Schirmers I test
   * Nausea, insomnia, headache, loss of appetite, malaise, diarrhoea and abdominal cramps may occur after herbal consumption

   Relatively few complications have been reported from the use of acupuncture. However, acupuncture can cause potentially serious side effects if not delivered properly by a qualified practitioner. The most common side effects after acupuncture include soreness, bruises, fatigue, lightheadedness and involuntary twitching of muscle. Should this event occur, increased frequency of visits to the eye clinic may be necessary.

   1.3.2 Potential Benefits There is no assurance participants will benefit from this study. However, their participation may contribute to the medical knowledge whether TCM medicine can fundamentally alter the pathological processes in dry eye. At the same time, regulatory bodies need to be reassured that TCM is safe in dry eye, so that more education and promotion of such treatment can benefit more people.
2. STUDY POPULATION 3.1 List The Number and Nature of Subjects to be Enrolled. One hundred and fifty eligible dry eye subjects will be screened and recruited from SCHMI.

3.2 Criteria for Recruitment and Recruitment Process

1. Subjects meet all the inclusion criteria listed below.
2. Clear of exclusion criteria.

Permission would be sought from the attending TCM physicians before subjects are being recruited. Eligible subjects will be counselled on the study. If subject is interested, informed written consent will be obtained from all participants. Thereafter, optometrsits at SCHMI will schedule a baseline visit to SERI for ocular monitoring.

3.3 Inclusion Criteria

For eligibility each participant presenting at SCHMI must be assessed by the TCM physician and optometrist, and found to satisfy every one of the following:

1. Age: 40-85 years, visual acuity better than logMAR of 1.0
2. Chief complaint should be dry eye
3. Symptoms:

   3.1. SPEED score > 6 3.2. TCM score satisfies lung-kidney yin deficiency profile
4. Signs:

4.1. TBUT (<10s) or Schirmer's test (<10mm/5 mins) 4.2 Any corneal fluorescein staining

3.4 Exclusion Criteria All subjects meeting any of the exclusion criteria at screening visit will be excluded from participation.

1. Glaucoma or other ophthalmic disease, eg. Extraocular muscle palsies, ectropion, entropion
2. Ocular allergies, eg. Allergic conjunctivitis, sinusitis, eczema, atopic keratoconjuntivitis
3. Known of thyroid disorders (diagnosed by physician)
4. Trichiasis
5. Eye surgeries patients including LASIK (within 1 year)
6. Steven-Johnson syndrome
7. Sjogren's syndrome
8. Eye related trauma (within 1 year)
9. Contact lens wear (within 1 year)
10. Punctal occlusion
11. Systemic disease requiring regular medication (except hypertension and lipidemia)
12. Pregnancy or planning to be pregnant
13. Requirement for medications such as anti-microbial, inflammatory, creams (except moisturizers or cosmetics), or steroidal therapies
14. Unable to do this clinical trial for any reason

4 STUDY DESIGN This is a randomized observer masked parallel group three arm interventional study.

Treatment arms

There will be 3 trial arms in this study:

* Control: Systane Ultra Eye drop (n=50)
* Systane Ultra Eye Drop and Acupuncture treatment (n=50)
* Systane Ultra Eye Drop and Herbs treatment (n=50)

Study duration: 5 Weeks Recruitment duration: 1 Year

4.1 Randomisation and Blinding

The randomisation procedure used will entail:

1. Presence of two witnesses
2. Drawing of lots
3. Randomization codes for the 3 groups will be noted. For e.g. 001A, 002B, 003C etc.
4. Study information related to randomisation will be filed and kept at SCHMI
5. Only unblinded personnel have access to the randomization code file

Randomisation will be done at SCHMI. Study members at SCHMI will be unblinded as they will be delivering TCM treatments to the subjects. However, study members at SERI will all be blinded so as to prevent unintentional biases when assessing and monitoring of ocular surface.

In a situation of a serious event, a decision on whether to open (break) the code for the specific patient is necessary. Although it is advantageous to retain the blind for all patients prior to final study analysis, when a serious adverse reaction is judged reportable on an expedited basis, it is recommended that the blind be broken only for that specific patient by the designated investigator who is unblind. It is also recommended that, when possible and appropriate, the blind be maintained for those persons, such as biometrics personnel, responsible for analysis and interpretation of results at the study's conclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-85 years, visual acuity better than logMAR of 1.0
2. Chief complaint should be dry eye
3. Symptoms:

   3.1. SPEED score > 6

   3.2. TCM score satisfies lung-kidney yin deficiency profile
4. Signs:

4.1. TBUT (<10s) or Schirmer's test (<10mm/5 mins) 4.2 Any corneal fluorescein staining

Exclusion Criteria:

1. Glaucoma or other ophthalmic disease, eg. Extraocular muscle palsies, ectropion, entropion
2. Ocular allergies, eg. Allergic conjunctivitis, sinusitis, eczema, atopic keratoconjuntivitis
3. Known of thyroid disorders (diagnosed by physician)
4. Trichiasis
5. Eye surgeries patients including LASIK (within 1 year)
6. Steven-Johnson syndrome
7. Sjogren's syndrome
8. Eye related trauma (within 1 year)
9. Contact lens wear (within 1 year)
10. Punctal occlusion
11. Systemic disease requiring regular medication (except hypertension and lipidemia)
12. Pregnancy or planning to be pregnant
13. Requirement for medications such as anti-microbial, inflammatory, creams (except moisturizers or cosmetics), or steroidal therapies
14. Unable to do this clinical trial for any reason

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in SPEED score (Week4-Week0) | 4 weeks
  Any improvement or discomfort in dry eye symptoms during 4 weeks

SECONDARY OUTCOMES:
Change in Tear Evaporimetry | 4 weeks
Change in TCM score (Lung-Kidney Yin deficiency) | 4 weeks
Change in Non Invasive Break Up Time | 4 weeks
Change in Schirmers I | 4 weeks
Change in Corneal fluorescein staining | 4 weeks
Change in Tear osmolarity | 4 weeks
Change in Tear meniscus height | 4 weeks
Change in Tear protein/ cytokine levels | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre/ Singapore Eye Research Institute, Singapore, Type A Choice Below ..., Singapore

REFERENCES:
- [Derived] Tong L, Htoon HM, Hou A, Acharya RU, Tan JH, Wei QP, Lim P. Acupuncture and herbal formulation compared with artificial tears alone: evaluation of dry eye symptoms and associated tests in randomised clinical trial. BMJ Open Ophthalmol. 2018 Jun 18;3(1):e000150. doi: 10.1136/bmjophth-2018-000150. eCollection 2018. PMID 30123846